CLINICAL TRIAL: NCT03198832
Title: Disease Periodontal Influence on Markers of Cardiovascular in Diabetes Mellitus Patients
Brief Title: oxLDL in Diabetes Mellitus Patients and Disease Periodontal
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Estadual Paulista Júlio de Mesquita Filho (Other)
Collaborators: LabviVale (Other)
Responsible Party: Principal Investigator, Maria Aparecida Neves Jardini, Professor, Universidade Estadual Paulista Júlio de Mesquita Filho
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CAAE:53785516.6.0000.0077
Record Dates: First submitted 2017-02-06; First posted 2017-06-26 (Actual); Last update posted 2018-11-14 (Actual); Status verified 2018-11

CONDITIONS: Type 2 Diabetes Mellitus With Periodontal Disease
Keywords: Periodontal Disease; Type 2 Diabetes Mellitus; Z-scan; Atherosclerosis
MeSH Terms: conditions — Periodontal Diseases; Diabetes Mellitus, Type 2; Atherosclerosis

STUDY DESIGN:
Intervention Model Description: Prospective double-blind controlled clinical study with a 6-month follow-up.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Type 2 diabetes mellitus and periodontitis (Sham Comparator): periodontal debridement in a single session.
  Interventions: Procedure: Non-surgical periodontal treatment
- Type 2 diabetes mellitus and without periodontitis (No Intervention): maintained every three months.

INTERVENTIONS:
Procedure: Non-surgical periodontal treatment — Debridement in a single session in which patients will be anesthetized and receive scaling and root planing with ultrasound equipment .
  Arms: Type 2 diabetes mellitus and periodontitis

SUMMARY:
Periodontal disease (PD) and diabetes mellitus type 2 (DM2) have the same inflammatory etiopathogenesis and demonstrate a bidirectional relationship, for DM2 affects the severity of PD, and this may contribute to the overall inflammatory burden of the individual, influencing the natural course DM2. The aim of this study is to establish whether individuals with DM with or without chronic periodontitis have an increase in oxLDL and what is the influence of periodontal treatment in the reduction of oxLDL with consequent improvement in Diabetes Mellitus parameters.

DETAILED DESCRIPTION:
Periodontal disease (PD) and diabetes mellitus type 2 (DM2) have the same inflammatory etiopathogenesis and demonstrate a bidirectional relationship, for DM2 affects the severity of PD, and this may contribute to the overall inflammatory burden of the individual, influencing the natural course DM2. The aim of this study is to establish whether individuals with DM with or without chronic periodontitis have an increase in oxLDL and what is the influence of periodontal treatment in the reduction of oxLDL with consequent improvement in Diabetes Mellitus parameters. 44 patients will be divided into 2 groups: Diabetic Patients with Chronic Periodontitis (DM2DP) and Diabetic Patients without Chronic Periodontitis (DM2). The DM2DP group will receive periodontal debridement and DM2 group will be treated with supragingival scaling. Both groups receive board control every 3 months. At baseline, 3 and 6 months after treatment, will be held making the clinical periodontal parameters (plaque index, gingival index, probing depth, gingival recession relative clinical attachment level and Periodontal Inflamed Surface Area (PISA) index) and blood collection for assessment serum inflammatory markers (oxLDL, LDL, HDL, total cholesterol, triglyceride, Interleukin (IL) IL-6, IL-8, IL-10, Tumor Necrosis Factor (TNF-α) and CRP). Biochemical analyzes will be carried out by Z-scan technique. The data obtained before and after periodontal therapy will be analyzed using the Shapiro-Wilk test.

ELIGIBILITY:
Inclusion Criteria:

* individuals older than 35 years with DM2 diagnosed for more than five years and HbA1c between 7% and 11%;
* be diagnosed with generalized chronic periodontitis: present at least 6 sites with periodontal pocket and loss of insertion above 5mm and two more bags with loss of insertion above 6mm;
* present at least 20 teeth;
* agree to participate in the study and sign the informed consent form

Exclusion Criteria:

* patients with cardiovascular diseases, cancer, gastrointestinal disorders, skin diseases, pregnancy, lactation, smoking, arthritis, lupus or other diseases of inflammatory origin;
* have undergone periodontal treatment in the last 12 months;
* have made use of antioxidant supplements, anti-inflammatories, or antibiotics within the previous 3 months;
* make use of medications that can alter the marking and concentration of oxLDL, for example, statins;
* have changed the medication for glycemic control in the last 3 months;
* present dental elements with pulpal or periapical inflammation.

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2016-05-02 (Actual); Primary Completion 2016-08-26 (Actual); Study Completion 2017-01-28 (Actual)

PRIMARY OUTCOMES:
Probing depth change | baseline, 90 and 180 days
  The change in the probing depth will be measure in millimeters before and after the treatment.

SECONDARY OUTCOMES:
oxLDL concentration Change | baseline and 180 days
  Change in concentration of oxLDL will be measured before and treatment.
LDL, HDL, Total cholesterol, Triacylglycerol | baseline and 180 days
  Blood concentration (g/ml) will be measured before and after periodontal therapy.
Plaque index | baseline, 90 and 180 days
  Number of teeth affected before and after periodontal treatment
Gingival index | baseline, 90 and 180 days
  number of teeth affected before and after periodontal treatment
Gingival Recession | baseline, 90 and 180 days
  Evaluated in millimeters before and after the treatment.
Clinical Attachment Level | baseline, 90 and 180 days
  Evaluated in millimeters before and after the treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Maria Jardini, PhD, Study Director — Universidade Estadual Paulista Julio de Mesquita Filho
Locations (1):
- São Jose Dos Campos, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No